CLINICAL TRIAL: NCT06439654
Title: Atlantic Lipid Lowering Treatment Optimization Program (ALLTOP): A Comprehensive Approach to the Treatment of Familial Hypercholesterolemia and Complex Dyslipidemias
Brief Title: Atlantic Lipid Lowering Treatment Optimization Program
Acronym: ALLTOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantic Health System (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Robert Fishberg, Principal Investigator, Atlantic Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2096455
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Familial Hypercholesterolemia; Lipoprotein Types--Lp System Lp(A) Hyperlipoproteinemia; Apolipoprotein B 100, Familial Defective; High Density Lipoprotein Deficiency; Low-Density-Lipoid-Type Hyperlipoproteinemia
Keywords: LDL-C; FH; complex dyslipidemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Lipoprotein Types--Lp System Lp(A) Hyperlipoproteinemia; Hypoalphalipoproteinemias | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: This is a prospective quantitative study of individuals with FH to examine the benefit of comprehensive supportive care to lower elevated LDL-C and sustain healthy levels through 36 months from baseline enrollment. We propose to demonstrate improvement in lipid parameters and outcomes in patients referred to the study. Specifically, we will target patients with documented hypercholesterolemia, hypertriglyceridemia, prior myocardial infarction, and personal or family history of coronary artery disease, who may be living with undiagnosed/untreated familial hypercholesterolemia FH.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LDL-C (Other): Most recent LDL-C result
  Interventions: Other: Supportive care

INTERVENTIONS:
Other: Supportive care — The study model will utilize the accepted standard of care while implementing key enhancements to proactively reach high-risk patients as early as possible. Wrap around comprehensive care is defined as database screening, outreach, encouraging genetic testing for participants and their family members, and provide ongoing education, medical management (e.g., adherence to FDA-approved medications), routine laboratory testing, specialist referrals, Epic referrals to integrated care support such as pharmacy, nutrition, social work, and community health), and routine follow-up either in-person or using virtual visits. Consultations with pharmacists, nutritionists and genetic counselors or specialists to manage co-morbidities may be requested.

SUMMARY:
Hypercholesterolemia is recognized as the major driver for cardiovascular morbidity and mortality. To help address this in our community, Atlantic Medical Group (AMG) formed a lipid workgroup chaired by Robert D. Fishberg, MD, and Jeffrey N. Feldman, MD. The overarching goal of the lipid workgroup is to enhance the treatment of lipid disorders in those patients with abnormal lipid levels by improving access to resources at the primary care practice level and specialty level. We aim to develop a model for primary and secondary prevention that integrates guidelines for treatment at the practice level. Our primary objective is to identify high-risk patients by utilizing the electronic health record and partnering with patients' primary care providers to provide comprehensive medical management.

DETAILED DESCRIPTION:
This study will screen patients with LDL-C >160 mg/dL and with evidence of familial hypertension, reach out (using secure chat) to the attending practitioner of such patients and inform the practitioner of our comprehensive services to address FH. A study team member will inform the practitioner that one of the study team plans to reach out to their patient to inform the patient of the study. Unless one of the study team receives notification by the practitioner that they want to opt out of this service for their patients, and do not want further interaction, the patient will be informed of the study and the consent process.

The research question is: Will an innovative comprehensive outreach approach, in conjunction with the primary care provider, reduce LDL-C levels in individuals with familial hypercholesteremia below individual baseline values, ideally at a level at or below 100 mg/dL.

ELIGIBILITY:
Inclusion Criteria:

* LDL-C ≥160 mg/dL
* Untreated LDL-C ≥190 with family history of CAD
* Prior MI and currently without optimized lipid-lowering therapy
* Family history of CAD in first degree relative
* Personal history of CAD
* Untreated triglycerides >500
* Elevated Lp(a) and/or high calcium scores
* Consenting individuals

Exclusion Criteria:

* Individuals who are pregnant
* Individuals who are incarcerated
* Individuals with a terminal illness
* Individuals who do not consent

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with LDL-C maintenance<100 | 6 months from enrollment in study
  LDL-C <100 mg/dL after at least six months of therapy

SECONDARY OUTCOMES:
Proportion of patients with LDL-C reaching <75 | 6 months from enrollment in study
  LDL-C <75 mg/DL
Proportion of patients with LDL-C reaching <55 | 6 months from enrollment in study
  LDL-C < 55mg/DL

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Fishberg, MD, Principal Investigator — Atlantic Health System
Locations (2):
- United States (2):
  - Atlantic Medical Group, Clark, New Jersey
  - Atlantic Medical Group, Springfield, New Jersey

IPD SHARING:
Plan to Share IPD: No
De-identified data will be disseminated in aggregate.

REFERENCES:
- [Background] Khera AV, Won HH, Peloso GM, Lawson KS, Bartz TM, Deng X, van Leeuwen EM, Natarajan P, Emdin CA, Bick AG, Morrison AC, Brody JA, Gupta N, Nomura A, Kessler T, Duga S, Bis JC, van Duijn CM, Cupples LA, Psaty B, Rader DJ, Danesh J, Schunkert H, McPherson R, Farrall M, Watkins H, Lander E, Wilson JG, Correa A, Boerwinkle E, Merlini PA, Ardissino D, Saleheen D, Gabriel S, Kathiresan S. Diagnostic Yield and Clinical Utility of Sequencing Familial Hypercholesterolemia Genes in Patients With Severe Hypercholesterolemia. J Am Coll Cardiol. 2016 Jun 7;67(22):2578-89. doi: 10.1016/j.jacc.2016.03.520. Epub 2016 Apr 3. PMID 27050191
- [Background] Amrock SM, Duell PB, Knickelbine T, Martin SS, O'Brien EC, Watson KE, Mitri J, Kindt I, Shrader P, Baum SJ, Hemphill LC, Ahmed CD, Andersen RL, Kullo IJ, McCann D, Larry JA, Murray MF, Fishberg R, Guyton JR, Wilemon K, Roe MT, Rader DJ, Ballantyne CM, Underberg JA, Thompson P, Duffy D, Linton MF, Shapiro MD, Moriarty PM, Knowles JW, Ahmad ZS. Health disparities among adult patients with a phenotypic diagnosis of familial hypercholesterolemia in the CASCADE-FH patient registry. Atherosclerosis. 2017 Dec;267:19-26. doi: 10.1016/j.atherosclerosis.2017.10.006. Epub 2017 Oct 6. PMID 29080546
- [Background] Kastelein JJ, Ginsberg HN, Langslet G, Hovingh GK, Ceska R, Dufour R, Blom D, Civeira F, Krempf M, Lorenzato C, Zhao J, Pordy R, Baccara-Dinet MT, Gipe DA, Geiger MJ, Farnier M. ODYSSEY FH I and FH II: 78 week results with alirocumab treatment in 735 patients with heterozygous familial hypercholesterolaemia. Eur Heart J. 2015 Nov 14;36(43):2996-3003. doi: 10.1093/eurheartj/ehv370. Epub 2015 Sep 1. PMID 26330422
- [Background] Alam L, Fishberg R, Echeverry T, Feldman J. Screening for familial hypercholesterolemia using Epic Secure Chat in comparison to Epic Letter as educational outreach. Journal of Clinical Lipidology. 2022;16(1):e20-e21. doi.org/10.1016/j.jacl.2021.09.029
- [Background] Writing Committee; Lloyd-Jones DM, Morris PB, Ballantyne CM, Birtcher KK, Covington AM, DePalma SM, Minissian MB, Orringer CE, Smith SC Jr, Waring AA, Wilkins JT. 2022 ACC Expert Consensus Decision Pathway on the Role of Nonstatin Therapies for LDL-Cholesterol Lowering in the Management of Atherosclerotic Cardiovascular Disease Risk: A Report of the American College of Cardiology Solution Set Oversight Committee. J Am Coll Cardiol. 2022 Oct 4;80(14):1366-1418. doi: 10.1016/j.jacc.2022.07.006. Epub 2022 Aug 25. No abstract available. PMID 36031461
- [Background] Myers KD, Farboodi N, Mwamburi M, Howard W, Staszak D, Gidding S, Baum SJ, Wilemon K, Rader DJ. Effect of Access to Prescribed PCSK9 Inhibitors on Cardiovascular Outcomes. Circ Cardiovasc Qual Outcomes. 2019 Aug;12(8):e005404. doi: 10.1161/CIRCOUTCOMES.118.005404. Epub 2019 Jul 23. PMID 31331194